CLINICAL TRIAL: NCT01734941
Title: A Phase 2 Randomized Three-Arm Double-Blind Placebo-Controlled Study to Evaluate the Safety and Efficacy of 16 Weeks of Treatment With Trichuris Suis Ova (TSO) Therapy in Pediatric Patients Ages 6 to 17 With Autism
Brief Title: TSO in Pediatric Autistic Spectrum Disorders
Acronym: TSO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Well tolerated but failed to demonstrate significant activity. So it did not meet its primary endpoint or key secondary endpoints.
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0522-12-HMO
Record Dates: First submitted 2012-11-19; First posted 2012-11-28 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2014-04

CONDITIONS: Autistic Spectrum Disorders
Keywords: Autism; Trichuris Suis Ova; Behavior; Irritability
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Behavior | interventions — Equipment and Supplies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TSO 2500 (Active Comparator): 2500 TSO every other week
  Interventions: Drug: TSO
- 7500 TSO (Active Comparator): 7500 TSO every other week
  Interventions: Drug: TSO
- Placebo (Placebo Comparator): placebo every other week.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TSO — There is evidence of a relationship between ASD symptomatology and immune dysfunction suggests that immunomodulatory treatments effective in other autoimmune disorders might be investigated in ASD, including Trichuris Ova Suis (TSO), a helminth porcine whipworm
  Other Names: Each dose of 2500 and 7500 active Trichuris suis ova will be provided; in 15 mL of aqueous suspension (supplied in 30 mL glass container); or matching placebo administered orally at the investigational center
  Arms: 7500 TSO; TSO 2500
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate and compare the safety and efficacy of Trichuris suis ova (TSO) therapy (versus placebo) in pediatric patients with autism.

Evaluation of the safety and tolerability of treatment with TSO in the target population across the dose range being tested is considered a primary objective, while the primary efficacy objective will be assessed via the change from baseline in the Aberrant Behavior Checklist (ABC) subscale scores.

Dose response will be considered a primary objective as well.

Secondary assessments of efficacy will be assessed via:

• The change from baseline in the Clinical Global Impression scale (CGI-I)

DETAILED DESCRIPTION:
This is a randomized, three-arm double-blind, placebo-controlled, single-center study to evaluate the effects of oral administration of Trichuris suis ova (as compared to placebo) in the treatment of pediatric patients diagnosed with Autism. The target sample size to be randomized into the study will be approximately 60, randomly assigned in a 1:1:1 ratio to one of three treatment groups:

1. Placebo (n= 20 patients). These patients will receive a blinded dose of placebo every other week.
2. 2500 TSO every other week (n= 20 patients). These patients will receive a blinded dose of TSO every other week
3. 7500 TSO every other week (n= 20 patients). These patients will receive a blinded dose of TSO every other week

Double-blind treatment will be given for a total of 16 weeks.

This study will have 3 phases:

* Screening period, comprising up to 5 weeks prior to Baseline (Day 1)
* Double-blind treatment period for 16 weeks
* An untreated follow-up period for 26 weeks. Following informed consent, patients will be screened on the basis of diagnosis of autism, vital signs, clinical laboratories medical history and a physical examination. Eligible patients will be randomized to double-blind treatment with TSO 2500 every other week, TSO 7500 every other week, or placebo every other week, in a ratio of 1:1:1. During the double-blind study phase, study drug will be provided in the clinic in a liquid form and will be administered every other week, starting with the Baseline visit, through Week 14. Week 14 is the last double-blind treatment administration of the study, while Week 16 is the primary time point for assessment of efficacy. Patients will return to the clinic every other week during the double blind treatment period.

After completion of the double-blind phase, patients will then return to the clinic 26 weeks following the last dose of study medication for a safety assessment and stool sample culture.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, ages 6 to 17 years, inclusive
2. Diagnosis via Diagnostic and Statistical Manual for Mental Disorders- Forth Edition (DSM-IV)-and confirmed by Autism Diagnostic Observation

   Schedule (ADOSI):
3. CGI-Severity score > 4 and ABC irritability score > 18
4. Mental age of > 18 months
5. Weight of at least ** kg
6. Currently psychotropic medication free or on stable dose of psychotropic medication for at least 3 months prior to the study.
7. Willing to comply with the schedule of study visits and protocol requirements
8. Patient and/or guardian have the ability to provide informed consent

Exclusion Criteria:

1. Previous diagnosis of Rett's Disorder, Aspergers Disorder, Childhood Disintegrative Disorder, Fragile X Syndrome, or other disorders on the autism spectrum
2. History of Bipolar Disorder, Psychotic Disorders, or major Depression
3. Seizure within the previous 6 months
4. Patient received antibiotic, antifungal or antiparasitic medication in the last 2 weeks prior to Screening and/or would potentially require this during the study treatment period
5. Patient with history of drug or alcohol abuse within 6 months prior to Screening
6. Patient with evidence of poor compliance with medical advice and instruction including diet or medication
7. Patient is unable or unwilling to swallow study medication suspension
8. Patient with a significant medical condition which puts the patient at risk for study participation and/or for any reason is considered by the Investigator to be an unsuitable candidate to receive TSO or is potentially put at risk by study procedures
9. Patient who has participated in another clinical trial within 30 days of Screening for this trial and/or any experimental treatment for this population
10. Females of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period
11. Females who are pregnant or breastfeeding at the time of enrollment
12. Patients with any of the following laboratory values:

    1. White blood cell count ≤ 3,000/mm3 (≤ 3.0 x 109/L) or ≥ 14,000/mm3 (≥14 x 109/L)
    2. Platelet count ≤ 100,000/μL (≤100 x 109/L)
    3. Serum creatinine ≥ 1.5 mg/dL (≥ 132.6 μmol/L) or >2 x upper limit of normal (ULN)
    4. AST (SGOT) or ALT (SGPT) > 2 x ULN
    5. Total bilirubin >2 mg/dL (34 μmol/L)
    6. Hemoglobin < 9 g/dL

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2014-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Aberrant Behavior Checklist (ABC) subscale scores | 16 weeks
  The ABC consists of 58 questions and the five subscales as described above. Each question on the ABC is rated on a 4-point scale: 0 = 'not a problem,' 1 ='the behavior is a problem but slight in degree,' 2 = 'the problem is moderately serious,' and 3 = 'the problem is severe in degree.' The subscale score is the sum of the responses to the questions that make up the subscale.

SECONDARY OUTCOMES:
Secondary assessments of efficacy will be assessed via: The change from baseline in the CY-BOCS, CGI-I, SRS, SCQ. | 49 weeks
  Secondary assessments of efficacy will be assessed via:
  • The change from baseline in the Clinical Global Impression - Improvement scale (CGI-I)

OTHER OUTCOMES:
Clinical Laboratory | 49 weeks
  Clinical laboratories will include hematology and serum chemistry panels, as well as C-reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Itai Berger, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- The Neuro-Cognitive Center, Pediatric Division, Hadassah-Hebrew University Medical Center, Jerusalem, Mount Scopus, Israel

REFERENCES:
- [Background] Summers RW, Elliott DE, Urban JF Jr, Thompson R, Weinstock JV. Trichuris suis therapy in Crohn's disease. Gut. 2005 Jan;54(1):87-90. doi: 10.1136/gut.2004.041749. PMID 15591509
- [Background] Fleming JO, Isaak A, Lee JE, Luzzio CC, Carrithers MD, Cook TD, Field AS, Boland J, Fabry Z. Probiotic helminth administration in relapsing-remitting multiple sclerosis: a phase 1 study. Mult Scler. 2011 Jun;17(6):743-54. doi: 10.1177/1352458511398054. Epub 2011 Mar 3. PMID 21372112